CLINICAL TRIAL: NCT06584851
Title: Evaluation of Microscopic Muscle Properties in Growing Children With Cerebral Palsy and Their Relation to Macroscopic Muscle Properties
Brief Title: 3D-Microscopic Muscle Architecture in Cerebral Palsy
Acronym: 3D-MMAP
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Desloovere, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S62645
Record Dates: First submitted 2024-05-24; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Spastic Cerebral Palsy
Keywords: Spastic cerebral palsy; Microscopic muscle properties; Muscle micro-biopsies; 3D freehand ultrasound; Histology; Cell culture; CP-phenotypes
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sonographically guided percutaneous needle micro-biopsies will be collected at the Medial Gastrocnemius and the Semitendinosus. Per biopsy, four muscle samples of +/- 20 mg will be collected per muscle on one location of the muscle, and useable for both histological and cell culture analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children with spastic cerebral palsy: Children between 2 and 9 years old.
- Typical developing children: Children between 2 and 9 years old.
- Adolescents and adults with HSP: Adolescents between 12 and 18 years of age and adults.
- Typically developing adolescents and adults: Age- and gender- matched with the recruited HSP patients

SUMMARY:
The focus of this study is to understand and define the mechanisms of the altered muscle development and growth on a microscopic level within a long-term perspective in children with cerebral palsy and to relate these findings to muscle macroscopic properties defined by muscle imaging, to neuromuscular symptoms and to treatment.

This study aims to (1) evaluate intrinsic microscopic muscle properties of young growing children with CP, and (2) to evaluate these muscle properties in relation to macroscopic properties, neuromuscular symptoms and to treatment.

Improved understanding of changes in microscopic muscle properties, and how they relate to macroscopic properties and to the neuromuscular symptoms as well as how they are influenced by treatment, has the potential to delineate CP phenotypes prone to intervention and to optimize treatment protocols or develop new treatments, leading to new avenues for improving function in CP.

The method to study microscopic muscle properties involves analysis of muscle biopsies (histological / immunohistochemistry analysis, SC and IC culture, gene expression). Biopsies will be collected using the minimally invasive percutaneous needle microbiopsy technique, suitable for collecting repeated samples over time in the same individual while still leading to sufficient tissue of good quality for subsequent analysis1,2. For the children with CP, the local hospital's tradition of applying general anesthesia for delivering BTX injections will be exploited to collect the muscle samples prior to the BTX session and the one-year follow-up, or general anesthesia planned for orthopedic surgery or diagnostic imaging such as MRI, etc. For the collection of the samples 3 months before the BTX session, as well as 3 months and 6 months after BTX injections, the common approach for microbiospy collection will be applied, with local sedation on the skin (Rapydan©) and fascia (Xylocaine©) and local anesthesia by using Kalinox© (nitrous oxide in oxygen) under supervision of the University Hospital PROSA team. Biopsies of TD muscles will be collected in children with no history of neurological disorder, nor musculoskeletal problems at the level of the gastrocnemius or semitendinosus, at the time of upper limb orthopedic or trauma surgery and thus always under general anesthesia. Ultrasound guided percutaneous muscle biopsy has been performed in children (2 months-18 years)3,4 and has proven to be safe and well-tolerated. A pilot study (S61110) was conducted to confirm that the microbiopsy technique is suitable for the analysis of microscopic muscle properties and is well-tolerated in children with CP.

Two specific research goals are planned, with hypotheses emerging from literature.

DETAILED DESCRIPTION:
Background:

Altered muscle properties in CP have been reported by our own as well as other research groups, macroscopically and microscopically. Hence, key experts in the field acknowledge that further progress in the understanding of the pathogenesis of altered muscle properties will be gained by performing studies that combine macro- and microscopic evaluations of muscle structures, to define different disease presentations. Previous research also showed that a variety of treatment modalities, such as muscle stretching, strengthening, or tone reduction, have beneficial effects on neuromuscular symptoms and on certain muscle properties. However, treatment outcomes are not always satisfying and seem to be muscle and patient-specific. Recent developments in instrumented assessment of these clinical symptoms highlighted their heterogeneity. By applying these novel instrumented assessments, we found that the emergence of different neuromuscular phenotypes was found, such as distinct classes of spasticity based on muscle activation patterns measured during passive stretches at different velocities. While our results highlight that these phenotypes react differently to treatment, their etiology remains unknown. These findings suggest that patient-specific treatment can be improved when tuned to more entirely defined phenotypes. A comprehensive description of the intrinsic muscle properties, including microscopic as well as macroscopic features, is an important next step to further delineate the phenotypes, such that they can support the clinical decision making.

The pathogenesis of altered muscle growth in CP children remains inconclusive. There is no doubt that mature muscles adapt in response to altered use patterns30, suggesting that hampered muscle growth is a secondary process. However, many studies were restricted to children older than 2 to 4 years, and are therefore unable to systematically address the etiology of muscle deformities31. There is an urgent need to study microscopic muscle properties in young children with CP, at different ages. Also, a complete longitudinal delineation of altered muscle growth, covering an extended malleable period of childhood, is still missing.

Moreover, therapy for children with CP in Western countries generally starts at a very young age and includes physiotherapy, stretching casts, orthoses and BTX injections, which are all directed at the muscle. The diverse treatment histories of the participants from previous studies most likely influenced the development of certain muscles. Of particular interest is treatment with BTX injections, which became a first-line CP therapeutic intervention to treat focal spasticity, by means of chemodenervation. While BTX treatment results in reduced muscle tone, increased joint Range Of Motion [ROM] and improved gait, an increasing number of publications have raised concern that BTX may compromise muscle growth. Human studies on microscopic properties post BTX are rare. So far, there are no in vitro studies on CP muscles that have investigated the direct action of BTX on adult muscle stem cells. This is actually needed, since stroke and CP patients are different (in age, growth impact and number of BTX sessions) and animal studies suggest different mechanisms of intramuscular changes post BTX between juvenile and mature muscles. Hence, there is an urgent need to thoroughly investigate the potential impact of BTX on muscle atrophy and integrity in CP using a prospective study design. Indeed, research and clinics could benefit from a more detailed and longitudinal analysis of muscle samples, where it would be possible to characterize the short- and long-term effects of BTX injections on muscle tissue and on muscle adult stem cells.

Furthermore, different mechanisms underlying the altered muscle growth may also interact. Whilst the diversity of phenotypes is likely to reflect the interplay of several factors, and different pathways have been suggested as presumed key players in the pathogenesis of altered muscle properties and neuromuscular symptoms, little understanding remains on the predominant effect in specific circumstances. Literature suggests a close interplay between the ECM and SCs, such that the composition and mechanical properties of the ECM regulate SC activity and renewal; and conversely, SCs dictate ECM composition. More CP-related research is necessary to determine the importance of alterations in SCs, ICs, and ECM components, and their interplay.

The etiology of CP may also be relevant to understand the pathogenesis of altered muscle properties.

Although prematurity and hypoxic-ischemic injury, placental insufficiency, and prenatal infection are well-recognized causes of CP, more than 30% of the children lack traditional risk factors. For many of these cases, a genetic base to their condition is suspected. Indeed, current estimates indicate that as many as 30% of CP cases may be genetic in nature. Hence, for at least part of the CP children, some muscle properties might also be genetically driven. Moreover, specific groups of patients with Hereditary Spastic Paraplegia (HSP) present with a very similar clinical picture as the bilaterally involved patients with CP (i.e. similar symptoms of spasticity, muscle weakness, reduced muscle control and altered muscle structure)

Aim:

Objective 1: To study MICROSCOPIC MUSCLE PROPERTIES in CP and define their onset at an early disease stage and their progress with growth and pathology, and to delineate their potential genetic nature (≈ WP 1).

Firstly, muscle biopsies will be collected to define microscopic properties of two age-groups of CP and TD children (2-5 versus 6-9 years). It is hypothesized that (1) a lower percentage of contractile material, increased collagen content, reduced number of SCs and altered fiber size distribution are observed in CP compared to TD children, and (2) these differences are age- and muscle-specific.

Secondly, since knowledge on early events and a follow-up of these events are lacking at the microscopic level, repeated biopsies will be collected in two CP groups (i.e. with and without BTX treatment history) , to study changes in the microscopic properties at different time-points pre- and post BTX injections. The microbiopsies under general anaesthesia (at the time of the BTX session and 1.2 year later, i.e. at the time of the repeated BTX-session), will be performed on the medial gastrocnemius and semitendinosus, while the microbiopsies under locale aneasthesia (at 3 months pre and 3 and 6 months post BTX) will be performed only on the medial gastrocnemius. It is hypothesized that (1) BTX-injection induce immediate altered structural muscle properties and molecular changes, which partly recover within 1.2 year, combined with (2) the trajectory of changes (such as collagen content and persistence of inflammatory cells) differs between BTX-naïve patients and patients with BTX treatment history, during the 1.2-year follow-up.

Thirdly, while literature suggests a close interplay between the ECM, SCs and ICs, there is a lack of CP-related research on the interaction between microscopic properties. A potential key regulatory factors that determine altered microscopic muscle properties will be defined, in particular, the relative importance of adult stem cell alterations by defining their interaction to ECM abnormalities. It is hypothesized that (1) the misbalanced interplay between adult stem cells and ECM is related to altered muscle properties, (2) the degree of misbalance evolves over time and (3) is muscle-specific.

Fouthly, recent literature suggests a genetic contribution to the pathology in about 30% of the children with CP, and subgroups of patients with HSP (SPG3a and SPG4) have identified genetic problems and present with similar clinical symptoms as the children with bilateral CP. This triggers a novel research pathway on the multi-lineage differentiation of induced pluripotent stem cells in a select group of patients with proven genetic mutation. It is hypothesized that that patient-specific cell modelling reflects genetic mutations, influencing the patient phenotype.

Objective 2: To delineate INTEGRATED CP PHENOTYPES prone to treatment, by identifying relations between different levels of muscle alterations (macro- and microscopic) and neuromuscular symptoms. The focus will be primarily on the symptom spasticity and on BTX treatment. (≈ WP 2).

Biopsy collection in the enrolled children of WP1 will always be preceded by ultrasound measures. As part of their routine clinical follow-up, these children also receive gait analysis and clinical assessments (using standard clinical scales) of neuromuscular symptoms before the treatment. Additionally, instrumented assessments of spasticity and strength will be performed. This allows integrated analysis on multiple datasets, to delineate integrated CP phenotypes. Firstly, relations between macro- and microscopic properties and spasticity will be explored. It is hypothesized that (1) macroscopic growth is significantly related to the number and behavior of SCs & ICs, to fiber type properties, and indirectly to ECM abnormalities, (2) the macroscopic parameter EI is associated to microscopic muscular tissue integrity, and (3) muscle properties are different between muscles classified by their spasticity patterns. Secondly, guidelines will be developed to fine-tune BTX treatment to the integrated phenotypes. It is hypothesized that (1) BTX induces altered muscle volume and integrity but does not change the number of SCs and (2) BTX response is significantly correlated to specific baseline CP phenotype markers (in particular to muscle integrity).

Methods/design:

To understand and define the mechanism and time course of muscle properties, different studies with different study designs will be applied. These studies are organized in two work packages, each covering one of the two specific research goals.

ELIGIBILITY:
CHILDREN WITH CP

Inclusion criteria

* Children (boys/girls) diagnosed with predominantly spastic type of CP
* Uni- or bilateral involvement
* Gross Motor Function Classification Scale (GMFCS) Level I-III50
* 2 to 9 years of age
* Planned for an orthopedic intervention that requires general anesthesia (botulinum toxin injections, orthopedic surgery, or diagnostic imaging such as Magnetic Resonance Imaging [MRI], etc.)

Exclusion criteria

* Presence of dystonia or ataxia
* Previous surgery less than 6 months at the investigated muscles
* Severe co-morbidities (that are likely to prevent proper assessment, such as severe cognitive problems)

TYPICALY DEVELOPING CHILDREN

Inclusion criteria

* Children (boys/girls)
* 2 to 9 years of age
* Planned for a surgical intervention that requires general anesthesia (pure pediatric upper limb orthopedic surgery or trauma surgery, or ophthalmic or ear-nose-throat surgery)

Exclusion criteria

* History of neurological problems
* History of orthopedic problems at the gastrocnemius or semitendinosus
* Trauma at the level of the lower limbs
* Involvement in an elite or high-performance sporting program (Children performing sports for > 3 5 hours/week will be excluded)

ADOSESCENTS WITH HSP of 12-18 years old and ADULTS WITH HPS

Inclusion criteria

* Adolescents (boys/girls) or adults (male/female) diagnosed with HSP, SPG3a or SPG4
* Gross Motor Function Classification Scale (GMFCS) Level I-III50
* Adolescents 12 to 18 years or adults 18-40 years of age

Exclusion criteria

* Presence of dystonia or ataxia
* Previous surgery less than 6 months at the investigated muscles
* Severe co-morbidities (that are likely to prevent proper assessment, such as severe cognitive problems)

TYPICALLY DEVELOPING ADOLESCENTS of 12-18 years old and HEALTHY ADULTS (age- and gender-matched with the recruited HSP patients)

Inclusion criteria

* Typically developing adolescents (boys/girls) and healthy adults (male/female), who are age and gender matched with the recruited HSP participants
* Adolescents 12-18 years of age or adults 18-40 years of age

Exclusion criteria

* History of neurological problems
* History of orthopedic or muscular problems at the gastrocnemius
* Trauma at the level of the lower limbs
* Involvement in an elite or high-performance sporting program (participants performing sports for > 5 hours/week will be excluded)
* Sport session less than 72 hours prior to the biopsy collection

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with spastic cerebral palsy, who have routine follow-up care at the CP reference center of the University Hospitals Leuven.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Muscle fiber size | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  Cross sectional area in µm of the fiber. Muscle fiber size will be assessed on cryosection stained with an antibody cocktail specific to laminin, myosin heavy chain (MHC)-I, MHC-IIA, MHC-IIB, MHC-embryonal and immunofluorescent detection will be done using appropriate secondary antibodies.
Muscle fibre type proportion | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  For each muscle, muscle fiber proportion will be assessed on cryosection stained with an antibody cocktail specific to laminin, myosin heavy chain (MHC)-I, MHC-IIA, MHC-IIB, MHC-embryonal and immunofluorescent detection will be done using appropriate secondary antibodies.
Capillary density | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  Capillaries /mm2 fiber and capillary to fiber ratio. Capillaries will be detected in-situ. Capillaries will be assessed using CD31 staining.
Satellite cell density | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  Number of satellite cells/mm2. Satellite cells will be detected in-situ. Co-localization of satellite cells will be assessed using Pax7 staining in conjunction with MHC-I/laminin, DAPI and CD31. Abundance of satellite cell content (Pax7+/DAPI+) will be counted and their association with the different fiber types will be identified.
Myogenic differentiation potential by means of fusion index for SC (satellite cells) | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  SCs will be isolated by Fluorescence-Activated Cell Sorting (FACs) based on the presence of surface markers CD56.Behaviour of SCs will be analysed using a cell proliferation assay and a myogenic or adipogenic differentiation assay.
Myogenic differentiation potential by means of fusion index for MABs (mesoangioblasts) | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  MABs will be isolated by Fluorescence-Activated Cell Sorting (FACs) based on the presence of surface markers ALP.
Overall change in muscle belly length of the medial gastrocnemius muscle and the semitendinosus muscle | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  Estimation of the muscle belly length by 3DfUS. Muscle volume will be normalized to anthropometric growth.
Overall change in muscle volume of the medial gastrocnemius muscle and the semitendinosus muscle | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  Estimation of the muscle belly volume by 3DfUS. Muscle volume will be normalized to anthropometric growth.
Overall changes in muscle activation patterns | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  Estimation of the muscle activation patterns using instrumented spasticity assessment.

SECONDARY OUTCOMES:
Overall changes in collagen content | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  Estimation of the collagen content (µg/mg) collected from a micro biopsy from the medial gastrocnemius muscle and the semitendinosus muscle.
Overall change in muscle composition of the medial gastrocnemius muscle and the semitendinosus muscle by means of echo-intensity | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  Muscle composition can be indirectly estimated based on echo-intensity. Echo-intensity represents the gray scale of the ultrasonography image and can be related to the muscle content of contractile and non-contractile elements. The echo-intensity is extracted and expressed on an 8bit gray scale in arbitrary units (the tones of a grayscale image with a bit depth of 8 ranges from 0 (black) to 255 (white) and all the 254 shades of gray in between).
Overall change in muscle tendon length of the medial gastrocnemius muscle and the semitendinosus muscle | Through a study participation of 1,2 years depending on the trajectory: 1 evaluation moment at baseline, 1 follow-up 1,2 years after, or 5 evaluations: 3 months pre, baseline, 3 months after, 6 months after and 1,2 years after baseline
  Through a study participation of 1,2 years, depending on the trajectory: one evaluation moment at baseline (BTX injection), or 1 evaluation moment extra 1,2 years after baseline (combined with a second BTX injection), or 5 evaluations 3 months pre baseline, baseline, 3 months after baseline, 6 months after baseline and 1,2 years after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, prof.dr., Principal Investigator — Department of Rehabilitation Sciences, KU Leuven, Belgium
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium